CLINICAL TRIAL: NCT04626921
Title: VISIONARY-MS LTE: A Multi-Center, Open-Label Long-Term Extension Study Assessing the Safety, Efficacy, Tolerability, and Pharmacokinetics of CNM-Au8 In Patients With Stable Relapsing Multiple Sclerosis
Brief Title: A Multi-Center, Open-Label Long-Term Extension Study of CNM-Au8 In Patients With Stable Relapsing Multiple Sclerosis
Acronym: VISIONMS-LTE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Clene Nanomedicine (Industry)
Collaborators: George Clinical (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNMAu8.201LTE
Record Dates: First submitted 2020-10-30; First posted 2020-11-13 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: MS; RMS; Multiple Sclerosis; Demyelination; Remyelination; Optic Neuropathy; Optic Neuritis; Gold; Nanocrystal; Multifocal VEP; Full Field VEP; Low contrast letter acuity
MeSH Terms: conditions — Multiple Sclerosis; Demyelinating Diseases; Optic Nerve Diseases; Optic Neuritis

STUDY DESIGN:
Intervention Model Description: Open-Label, Long-Term Extension.
Masking Description: None, open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active treatment with 30 mg of CNM-Au8 (Experimental): Highly pure elemental Au nanocrystals are suspended in deionized water buffered with 0.546 mg/mL (6.5 mM) sodium bicarbonate (NaHCO3) concentrated up to 0.5 mg/mL (500 ppm) Au.
  Interventions: Drug: CNM-Au8

INTERVENTIONS:
Drug: CNM-Au8 — 30 mg of CNM-Au8

SUMMARY:
Open-label, long-term extension study available to participants who have completed CNMAu8.201.

DETAILED DESCRIPTION:
This open-label, long-term extension study is only available to participants who have completed CNMAu8.201 (VISIONARY-MS). The Week 48/End-of-Study Visit for study CNMAu8.201 (VISIONARY-MS) will serve to establish the Baseline for electrophysiological, functional, morphological vision testing, as well as the neurological and outcome assessments. Participants will receive open-label CNM-Au8 throughout the study. All participants will receive a daily dose of 30 mg CNM-Au8 for the entire open-label, long-term extension study. The dose for participants may be adjusted once efficacy and safety data from study CNMAu8.201 becomes available, which may occur after participants have already started this study. Based upon a review of data and Sponsor or PI recommendation, this open-label, long-term extension study may be discontinued once each participant reaches her/his 48-week visit.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have completed study CNMAu8.201.
* Able to understand and give written informed consent.

Exclusion Criteria:

* Lack of treatment compliance during participation in the CNMAu8.201 (VISIONARY-MS) study.
* Positive pregnancy test.
* Any history of previous malignancy, with the exception of basal cell carcinoma of the skin or in situ carcinoma of the cervix, post documented full resections, with clean margins.
* Based on the Investigator's judgment, any concurrent chronic or acute illness or unstable medical condition that could confound the results of safety assessments, increase risk to the participant, or lead to difficulty complying with the protocol; any untreated or unstable psychiatric disease including depression, bipolar and psychosis.
* Participant is considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt, or is currently demonstrating active suicidal ideation.

Following clinical and serology sample analysis conducted at the end-of-study visit for CNMAu8.201 (VISIONARY-MS), participants may be removed from this long term extension study if any of the following criteria are met, at the discretion of the Medical Monitor and/or Sponsor's Medical Representative:

* Positive serology for viral hepatitis B and/or C and/or human immunodeficiency virus (HIV).
* Abnormal liver function tests (aspartate aminotransferase [ASAT] or alanine aminotransferase [ALAT] > 2x upper limit of normal range (ULN) or total bilirubin > 2x ULN or alkaline phosphatase (AP) > 3x ULN).
* Participants with clinically significant hepatic or renal dysfunction or clinical laboratory findings that would limit the interpretability of change in liver or kidney function (e.g., glomerular filtration rate < 40 mL/min [based on creatinine clearance according to Cockcroft-Gault equation]), or those with low platelet counts (<150 x 109 per liter) or eosinophilia (absolute eosinophil count of ≥500 eosinophils per microliter) at the EOS visit for CNMAu8.201 (Visionary-MS).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Change in Best-Corrected Low-Contrast Letter Acuity score. | 2 years
  Mean change in BC-LCLA from baseline to end of study across all eyes as measured by 2.5% low contrast Sloan Letter Chart.
Incidence of treatment-emergent AEs throughout the study. | 2 years
  Safety endpoint include incidence of treatment-emergent AEs.

SECONDARY OUTCOMES:
Measure of neurological function assessed by a functional composite responder analysis. | 2 years
  Mean change in Functional Composite Responder Analysis Score from Baseline to End of Study.

OTHER OUTCOMES:
Change in best corrected Low-Contrast Letter Acuity score for total number of correct letter. | 2 years
  BC-LCLA score is the sum of all correctly identified letters up to the last line on the 2.5% Sloan Chart able in which three (3) or more letters are correctly read plus all correct letters on the following line. Scale is 70 - 0 with 70 being able to see all letters, 0 was unable to read any letters.
Change in Best Corrected High Contrast Visual Acuity | 2 years
  Mean change from Baseline in best-corrected high contrast visual acuity (BCHCVA), as measured by EDTRS in the affected and fellow eye. Scale is 70 - 0 with 70 being able to see all letters, 0 was unable to read any letters.
VEP latency for Multi-Focal visual evoked potential. | 2 years
  Mean change in average mf-VEP latency for the affected eye from the average Baseline mf-VEP latency of the affected eye.
VEP latency for Full Field Visual Evoked Potential | 2 years
  Mean change in average ff-VEP latency for the affected eye from the average Baseline ff-VEP latency of the affected eye.
VEP Amplitude for Multi-Focal Visual Evoked Potential | 2 years
  Mean change in average amplitude for the affected eye from the average Baseline of the affected eye (for all measurable segments).
VEP Amplitude for Full Field Visual Evoked Potential | 2 years
  Mean change in average amplitude for the affected eye from the average Baseline of the affected eye (for all measurable segments).
OCT of the Retinal Nerve Fiber Layer (RNFL) by Peripapillary Scan | 2 years
  Percentage change in average thicknesses of the RNFL for the affected eye and the fellow eye from their respective Baselines.
OCT of the Retinal Layers by Macular Scan evaluating Ganglion cell and inner plexiform. | 2 years
  Percentage change in mean thicknesses of the GCIP for the affected eye and the fellow eye from their respective Baselines as determined by segmentation of SD-OCT.
OCT of the Retinal Layers by Macular Scan evaluating Ganglion cell layer. | 2 years
  Percentage change in mean thicknesses of the GCL for the affected eye and the fellow eye from their respective Baselines as determined by segmentation of SD-OCT.
OCT of the Retinal Layers by Macular Scan evaluating Inner nuclear layer. | 2 years
  Percentage change in mean thicknesses of the inner nuclear layer for the affected eye and the fellow eye from their respective Baselines as determined by segmentation of SD-OCT.
OCT of the Retinal Layers by Macular Scan evaluating outer nuclear layer. | 2 years
  Percentage change in mean thicknesses of the outer nuclear layer for the affected eye and the fellow eye from their respective Baselines as determined by segmentation of SD-OCT.
MRI Evaluation of the Mean change in whole brain and OR T2 lesion volume. | 2 years
  Mean change in whole brain and OR T2 lesion volume from Baseline
MRI Evaluation of the Mean change in whole brain and optic radiation T1 hypo-intense lesion volume. | 2 years
  Mean change in whole brain and optic radiation T1 hypointense lesion volume from Baseline.
MRI Evaluation of the Proportion of Baseline Gd+ lesions converting to black holes. | 2 years
  Proportion of Baseline Gd+ lesions converting to black holes.
MRI Evaluation of the Volume of Baseline Gd+ lesions converting to T1 hypointense lesions. | 2 years
  Volume of Baseline Gd+ lesions converting to T1 hypointense lesions.
MRI Evaluation of the Mean percent whole brain volume change (PBVC) from baseline. | 2 years
  Mean percent whole brain volume change (PBVC) from baseline.
MRI Evaluation of the Mean Percent Cerebral Cortical Change from Baseline | 2 years
  Mean Percent Cerebral Cortical Change from Baseline
MRI Evaluation of the Mean Percent Thalamic Volume Change from Baseline. | 2 years
  Mean Percent Thalamic Volume Change from Baseline.
MRI Evaluation of the Mean Percent Deep Grey Nuclei Volume Change from Baseline. | 2 years
  Mean Percent Deep Grey Nuclei Volume Change from Baseline
MRI Evaluation of the Mean change in number of whole brain new/enlarging T2 lesion(s) from baseline. | 2 years
  Mean change in number of whole brain new/enlarging T2 lesion(s) from baseline.
Mean change in whole brain DTI/MTR from baseline. | 2 years
  DTI- Diffusion Tensor Imaging, MTR- Magnetization Transfer Ratio.
Mean change in optic radiation lesional/non-lesional fibre DTI / MTR difference from Baseline (fiber based, individually reported for each baseline OR lesion). | 2 years
  Individual OR lesion MRI analysis
Mean change in MWF from Baseline in the whole brain. | 2 years
  Myelin Water Fraction MRI Analysis

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Sydney Brain Mind Centre, Camperdown, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Menzies Institute for Medical Research, Hobart, TAZ
  - The Alfred Centre Department of Neuroscience, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No